CLINICAL TRIAL: NCT07288489
Title: A Phase 3 Prospective Randomised Clinical Trial of VMX-C001 vs Usual Pharmacological Care in Patients Receiving a FXa Direct Oral Anticoagulant (FXa DOAC) Who Require Urgent Surgery or Other Invasive Procedure That is Associated With a High Risk of Bleeding, With or Without Planned Administration of Heparin (EQUILIBRIX-S)
Brief Title: Phase 3 Trial of VMX-C001 vs Usual Pharmacological Care in Patients Taking a FXa Direct Oral Anticoagulant Who Require Urgent Surgery With or Without Heparin.
Acronym: EQUILIBRIX-S
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VarmX B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMX-C001-06
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Blood Loss, Surgical; Coagulation Disorder
Keywords: Direct oral anticoagulant (DOAC); Human coagulation factor; Surgery
MeSH Terms: conditions — Blood Loss, Surgical; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VMX-C001 (Experimental): Participants will be administered VMX-C001 before undergoing the required procedure.
  Interventions: Drug: VMX-C001
- Usual Pharmacological Care (Active Comparator): Participants will be given the usual treatment used by the site for patients receiving FXa DOACs when undergoing the required procedure.
  Interventions: Drug: Usual Pharmacological Care

INTERVENTIONS:
Drug: VMX-C001 — VMX-C001 will be administered prior to commencement of procedure.
  Arms: VMX-C001
Drug: Usual Pharmacological Care — Usual pharmacological care should be treatment planned to restore coagulation or support haemostasis for the required procedure.
  Arms: Usual Pharmacological Care

SUMMARY:
The goal of this clinical trial is to learn if VMX-C001 works to to allow blood clotting control in participants who take FXa Direct Oral Anticoagulants (DOACs) during surgery or other invasive procedures that carry a high risk of bleeding. The main question it aims to answer is:

● What is the proportion of participants in whom the stopping of bleeding was classed as good or excellent during the procedure, as judged by a group of experts who did not know which treatment was given?

Researchers will compare VMX-C001 to the usual treatment that would be given for the required procedure.

Participants will:

* Be given either VMX-C001 or usual treatment before they undergo the required procedure in theatre
* Have regular clinical assessments, including laboratory tests, during their hospital stay following the procedure
* Return to the clinic for a check-up and tests approximately 28 days after the procedure was conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged ≥18 years.
2. The patient or legally authorised representative (LAR) has given written informed consent.
3. The patient requires urgent surgery/procedure for which the risk of bleeding is considered high and for which haemostasis is considered necessary.
4. The patient has a significant FXa DOAC level at the time of procedure.
5. The patient would require treatment (usual pharmacological care) to restore coagulation for the required procedure.
6. The patient must be willing to use appropriate contraception.

Exclusion Criteria:

1. The patient is known for any reason, other than administration of a FXa DOAC, to have an increased risk of bleeding compared to a patient in a similar clinical situation.
2. The patient has received any non FXa DOAC anticoagulants within 7 days of Screening or has received heparin (UFH or LMWH) within 3 days of Screening.
3. The patient has received any of the prespecified medications not allowed in the 7 days prior to Randomisation.
4. The patient was treated with an investigational drug <30 days or 5 half-lives, whichever is longer, prior to Screening.
5. Expected survival, in the Investigator's judgement, is <3 months due to comorbidity.
6. Patients in whom the Investigator considers it is not possible to estimate the expected blood loss.
7. Known "Do Not Resuscitate" order or similar advanced directive.
8. Cardiogenic shock at the time of screening unless related to the need for the required procedure.
9. The patient has sepsis (including severe sepsis or septic shock) at the time of screening.
10. The patient is pregnant or a lactating female.
11. Known hypersensitivity to any component of VMX-C001 or hamster proteins.
12. Patients who, in the opinion of the Investigator, should not participate in the study for any other reason, or inability to comply with the protocol.
13. Prior exposure to VMX-C001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Effect of VMX-C001 versus usual pharmacological care on haemostasis | From start to end of required procedure (Day 1).
  Proportion of participants with good or excellent haemostatic efficacy during the required procedure.

SECONDARY OUTCOMES:
Effect of VMX-C001 versus usual pharmacological care on FXa DOAC induced anticoagulation measured by dilute prothrombin time (dPT). | From Pre-procedure assessment compared to baseline (Randomisation) (Day 1).
  Change in dPT.
Effect of VMX-C001 versus usual pharmacological care on FXa DOAC induced anticoagulation as measured by dilute Russell Viper Venom Time (dRVVT). | From Pre-procedure assessment compared to baseline (Randomisation) (Day 1).
  Change in dRVVT.
Effect of VMX-C001 versus usual pharmacological care on the extent of actual blood loss compared to expected blood loss during procedure. | From start to end of required procedure (Day 1).
  Percentage of expected blood loss.
Effect of VMX-C001 versus usual pharmacological care on bleeding severity. | Start of procedure (Day 1).
  Bleeding severity at the Start of procedure using a 5 point scale (grades 0 [no bleeding] to 4 [life threatening])
Effect of VMX-C001 versus usual pharmacological care on bleeding severity prior to procedure. | Between Randomisation and Pre-procedure timepoint (Day 1).
  Bleeding severity measured by blood loss.

CONTACTS AND LOCATIONS:
Locations (26):
- United States (16):
  - Chandler Regional Medical Center (CRMC), Chandler, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth John C Lincoln Medical Center, Phoenix, Arizona
  - Stanford Hospital and Clinics, Stanford, California
  - Denver Metro Orthopedics, P.C. - Englewood Location, Englewood, Colorado
  - Medical Center of the Rockies, Fort Collins, Colorado
  - Christiana Care, Newark, Delaware
  - University of South Florida, Tampa, Florida
  - University of Iowa Health Care, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beaumont Hospital, Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy Campus, Troy, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Texas Tech University Health Sciences Center - El Paso, El Paso, Texas
  - The University of Texas McGovern Medical School at Houston, Houston, Texas
- Australia (6):
  - Royal Brisbane and Women's Hospital (RBWH), Herston, Queensland
  - Mater Private Hospital, South Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - St Vincent Hospital, Melbourne, Fitzroy, Victoria
  - Alfred Health, Melbourne, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- New Zealand (4):
  - Auckland City Hospital, Grafton, Auckand
  - Aotearoa Clinical Trials - Middlemore (ACTT) Middlemore Hospital, Papatoetoe, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
  - Wellington Hospital, Newtown, Wellington Region

IPD SHARING:
Plan to Share IPD: Undecided